CLINICAL TRIAL: NCT03821155
Title: Which Treatment is Most Effective When Treating Vestibular Neuritis: Corticosteroid Treatment Alone or Combined Corticosteroid Treatment and Vestibular Rehabilitation?
Brief Title: Does Vestibular Rehabilitation Significantly Improve the Level of Vestibular Function Following Vestibular Neuritis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Dan Dupont Hougaard, MD, Assistant Professor, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-166
Record Dates: First submitted 2019-01-21; First posted 2019-01-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Vestibular Neuritis
Keywords: Vestibular Neuritis; SHIMP (suppressing head impulse paradigm); SVV (subjective visual vertical); Vestibular rehabilitation; Prednisolone; v-HIT (video head impulse test); Vestibular Neuronitis
MeSH Terms: conditions — Vestibular Neuronitis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Intervention Model Description: Patients randomized to two different treatments:
  1. corticosteroid treatment ("prednisolone")
  2. combined corticosteroid treatment ("prednisolone") and vestibular rehabilitation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuritis vestibularis (group 1) (Active Comparator): Corticosteroid ("prednisolone")
  Interventions: Drug: Corticosteroid
- Neuritis vestibularis (group 2) (Experimental): Corticosteroid ("prednisolone") + vestibular rehabilitation
  Interventions: Other: Vestibular rehabilitation; Drug: Corticosteroid

INTERVENTIONS:
Other: Vestibular rehabilitation — Specialized physical therapy aimed at restoring balance
  Arms: Neuritis vestibularis (group 2)
Drug: Corticosteroid — Prednisolone

SUMMARY:
To investigate which treatment option (corticosteroid treatment alone or combined corticosteroid treatment and vestibular rehabilitation) is the most effective in patients diagnosed with vestibular neuritis.

DETAILED DESCRIPTION:
Patients diagnosed with vestibular neuritis will we consider for enrollment. Each patient will undergo randomization for a specific treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years of age
2. Medical history compatible with vestibular neuritis
3. Verification of vestibular neuritis with positive romberg test, pathological v-HIT and horizontal nystagmus with a rotatory component.

Exclusion Criteria:

1. Former medical history with vestibular dysfunction
2. Medical history or objective signs of cochlear dysfunction before, during or after onset of vestibular neuritis
3. Onset of symptoms 14 days before recruitment to the study
4. Focal neurological symptoms/signs
5. Contraindication to prednisolone treatment
6. Problem with participating in vestibular rehabilitation due to muscular-skeletal disease ect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Suppressing head impulse paradigm (SHIMP) | 6 month
  SHIMP equipment will objectively quantify change of vestibular function.
Subjective visual vertical (SVV) | 6 month
  SVV test will objectively quantify the experienced spatial orientation as an indicator of visual and vestibular otolithic function
Video head impulse test (v-HIT) | 6 month
  v-HIT equipment will objectively quantify change of vestibular function.
Dizziness handicap inventory (DHI) questionnaire | 6 month
  Fulfillment of the questionnaire "Dizziness Handicap Inventory" (DHI) will quantify the level of experienced vertigo.

CONTACTS AND LOCATIONS:
Overall Officials: Dan D Hougaard, MD, Principal Investigator — Aalborg University Hospital; Martin H Wolder, MS, Principal Investigator — Aalborg University Hospital
Locations (1):
- Department of Otolaryngology, Head & Neck Surgery and Audiology, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No